CLINICAL TRIAL: NCT01283971
Title: A Randomized, Open-label, Parallel-group Study of the Reduction of Signs and Symptoms During Treatment With Tocilizumab Versus Adalimumab, Both in Combination With MTX, in Patients With Moderate to Severe Active Rheumatoid Arthritis and an Inadequate Response to Treatment With Only One TNF Inhibitor
Brief Title: A Study of RoActemra/Actemra (Tocilizumab) Versus Adalimumab in Combination With Methotrexate (MTX) in Patients With Moderate to Severe Active Rheumatoid Arthritis And an Inadequate Response to Treatment With Only One Tumor Necrosis Factor (TNF)-Inhibitor
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: The study was closed due to the slow enrollment rate.
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MA25522; 2010-023587-40 (EudraCT Number)
Record Dates: First submitted 2011-01-25; First posted 2011-01-26 (Estimated); Results first posted 2014-02-10 (Estimated); Last update posted 2014-02-10 (Estimated); Status verified 2014-01

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — tocilizumab; Adalimumab; Methotrexate; Folic Acid

ARMS (2):
- Tocilizumab + Methotrexate (Experimental): Tocilizumab 8 mg/kg intravenous (IV) every 4 weeks + Placebo to adalimumab subcutaneous (SC) every 2 weeks for 24 weeks. All participants received methotrexate 10-25 mg and folate at least 5 mg/kg weekly.
  Interventions: Drug: tocilizumab [RoActemra/Actemra]; Drug: placebo to adalimumab; Drug: methotrexate; Drug: folate
- Adalimumab + Methotrexate (Active Comparator): Adalimumab 40 mg SC every 2 weeks + Placebo to tocilizumab IV every 4 weeks for 24 weeks. All participants received methotrexate 10-25 mg and folate at least 5 mg/kg weekly.
  Interventions: Drug: adalimumab; Drug: placebo to tocilizumab; Drug: methotrexate; Drug: folate

INTERVENTIONS:
Drug: tocilizumab [RoActemra/Actemra] — Tocilizumab 8 mg/kg IV every 4 weeks for 24 weeks.
  Other Names: RoActemra/Actemra
  Arms: Tocilizumab + Methotrexate
Drug: adalimumab — Adalimumab 40 mg SC every 2 weeks.
  Arms: Adalimumab + Methotrexate
Drug: placebo to tocilizumab — Placebo to tocilizumab IV every 4 weeks for 24 weeks.
  Arms: Adalimumab + Methotrexate
Drug: placebo to adalimumab — Placebo to adalimumab SC every 2 weeks for 24 weeks.
  Arms: Tocilizumab + Methotrexate
Drug: methotrexate — Methotrexate 10-25 mg weekly.
Drug: folate — Folate at least 5 mg weekly.

SUMMARY:
This randomized, parallel-group study will assess the efficacy and safety of RoActemra/Actemra (tocilizumab) versus adalimumab, both in combination with methotrexate (MTX) in patients with moderate to severe active rheumatoid arthritis. Patients, already treated with MTX at stable doses, will be randomized to receive either RoActemra/Actemra 8 mg/kg intravenously (IV) every 4 weeks or adalimumab 40 mg subcutaneous (SC) every 2 weeks. All patients will receive methotrexate (10-25 mg weekly) and folate (at least 5 mg weekly). The anticipated time on study treatment is 24 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients, >/= 18 years of age
* Rheumatoid arthritis of >/= 6 months duration (according to American College of Rheumatology (ACR) criteria)(according to ACR criteria)
* Inadequate response due to inefficacy of treatment (for at least 3 months) with only one approved Tumor Necrosis Factor (TNF)-agent other than adalimumab Depending on the TNF-inhibitor, last dose of TNF-inhibitor should have been 1 to 8 weeks before randomization to the study
* On methotrexate treatment for >/=12 weeks immediately prior to baseline, with stable dose (10-25 mg/week) for the last 8 weeks
* Disease Activity Score (DAS28) >3.2 at baseline
* Oral corticosteroids (</=10 mg/day prednisone or equivalent) and non-steroidal anti-inflammatory drugs (NSAIDs) are permitted if the dose has been stable for >/=6 weeks prior to baseline.

Exclusion Criteria:

* Major surgery (including joint surgery) within 8 weeks prior to screening or planned surgery within 6 months following randomization
* Rheumatic autoimmune disease other than rheumatoid arthritis
* Prior history of or current inflammatory joint disease other than rheumatoid arthritis
* Functional class IV (ACR criteria)
* History of severe allergic reaction to human, humanized or murine monoclonal antibodies
* Known active current or history of recurrent infection (including tuberculosis)
* Primary or secondary immunodeficiency (history of or currently active)
* Body weight >150 kg
* Previous treatment with any cell-depleting therapies
* Previous treatment with tocilizumab
* Intra-articular or parenteral corticosteroids within 6 weeks prior to baseline.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2011-05; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (158):
- United States (98):
  - Huntsville, Alabama
  - Phoenix, Arizona
  - Tucson, Arizona
  - Covina, California
  - Escondido, California
  - Huntington Beach, California
  - La Mesa, California
  - Lakewood, California
  - Long Beach, California
  - Los Angeles, California
  - Sacramento, California
  - San Diego, California
  - Westlake Village, California
  - Whittier, California
  - Bridgeport, Connecticut
  - Hamden, Connecticut
  - Norwich, Connecticut
  - Newark, Delaware
  - Aventura, Florida
  - Fort Lauderdale, Florida
  - Jupiter, Florida
  - Melbourne, Florida
  - Naples, Florida
  - Ocala, Florida
  - Orlando, Florida
  - Ormond Beach, Florida
  - Palm Habor, Florida
  - Palm Harbor, Florida
  - Sarasota, Florida
  - Tamarac, Florida
  - Tampa, Florida
  - Atlanta, Georgia
  - Valdosta, Georgia
  - Idaho Falls, Idaho
  - Chicago, Illinois
  - Maywood, Illinois
  - Moline, Illinois
  - Springfield, Illinois
  - Fort Wayne, Indiana
  - South Bend, Indiana
  - Lexington, Kentucky
  - Baton Rouge, Louisiana
  - Monroe, Louisiana
  - Annapolis, Maryland
  - Cumberland, Maryland
  - Frederick, Maryland
  - Hagerstown, Maryland
  - Fall River, Massachusetts
  - Worcester, Massachusetts
  - Battle Creek, Michigan
  - Lansing, Michigan
  - Petoskey, Michigan
  - Saint Claire Shores, Michigan
  - Biloxi, Mississippi
  - Flowood, Mississippi
  - Tupelo, Mississippi
  - Springfield, Missouri
  - St Louis, Missouri
  - Reno, Nevada
  - Clifton, New Jersey
  - Manalapan, New Jersey
  - New Brunswick, New Jersey
  - Brooklyn, New York
  - New York, New York
  - Syracuse, New York
  - Charlotte, North Carolina
  - Greensboro, North Carolina
  - Greenville, North Carolina
  - Raleigh, North Carolina
  - Washington, North Carolina
  - Cleveland, Ohio
  - Middleburg Heights, Ohio
  - Toledo, Ohio
  - Oklahoma City, Oklahoma
  - Lake Oswego, Oregon
  - Duncansville, Pennsylvania
  - Philadelphia, Pennsylvania
  - Pittsburgh, Pennsylvania
  - Willow Grove, Pennsylvania
  - Wynnewood, Pennsylvania
  - Wyomissing, Pennsylvania
  - Charleston, South Carolina
  - Myrtle Beach, South Carolina
  - Jackson, Tennessee
  - Memphis, Tennessee
  - Austin, Texas
  - Carrollton, Texas
  - Corpus Christi, Texas
  - Houston, Texas
  - Mesquite, Texas
  - San Antonio, Texas
  - Sugar Land, Texas
  - Arlington, Virginia
  - Kennewick, Washington
  - Spokane, Washington
  - Tacoma, Washington
  - Clarksburg, West Virginia
  - Franklin, Wisconsin
- Denmark (3):
  - Aalborg
  - Elsinore
  - Silkeborg
- Finland (3):
  - Helsinki
  - Hyvinkää
  - Jyväskylä
- France (10):
  - Grenoble
  - Lille
  - Limoges
  - Metz
  - Montpellier
  - Mulhouse
  - Nantes
  - Orléans
  - Paris
  - Toulouse
- Germany (16):
  - Berlin
  - Düsseldorf
  - Erfurt
  - Erlangen
  - Frankfurt am Main
  - Gommern
  - Hamburg
  - Hanover
  - Heidelberg
  - Herne
  - Hildesheim
  - München
  - Osnabrück
  - Regensburg
  - Rostock
  - Tübingen
- Greece (3):
  - Athens
  - Heraklion
  - Thessaloniki
- Italy (5):
  - Florence
  - Milan
  - Pavia
  - Pisa
  - Roma
- Nijmegen, Netherlands
- Caguas, Puerto Rico
- Russia (4):
  - Kemerovo
  - Moscow
  - Ufa
  - Ulyanovsk
- Spain (8):
  - Sabadell, Barcelona
  - A Coruña, La Coruña
  - Santiago de Compostela, La Coruña
  - Madrid, Madrid
  - Málaga, Malaga
  - Oviedo, Principality of Asturias
  - Valenica, Valencia
  - Barakaldo, Vizcaya
- Sweden (6):
  - Gothenburg
  - Huddinge
  - Lund
  - Malmo
  - Umeå
  - Västerås

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Adalimumab + Methotrexate | Tocilizumab + Methotrexate
Started | 48 | 48
Intent to Treat Population | 46 | 48
Completed | 33 | 36
Not Completed | 15 | 12
Not completed — Adverse Event | 3 | 5
Not completed — Insufficient therapeutic responses | 3 | 3
Not completed — Protocol Violation | 5 | 1
Not completed — Refused treatment | 3 | 1
Not completed — Failure to return | 0 | 1
Not completed — Administrative reasons | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Adalimumab + Methotrexate | Tocilizumab + Methotrexate | Total
Number analyzed (Participants) | 48 | 48 | 96
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.3 (11.89) | 51.3 (12.51) | 52.8 (12.2)
Age, Customized [Number; unit: Participants]
  <50 years | 16 | 20 | 36
  50 to 64 years | 22 | 18 | 40
  ≥65 to 75 years | 9 | 10 | 19
  >75 years | 1 | 0 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40 | 38 | 78
  Male | 8 | 10 | 18

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Disease Activity Score 28 Joints (DAS28) Remission at Week 24
Description: The DAS28 score is a measure of the patient's disease activity calculated using the tender joint count (TJC) [28 joints], swollen joint count (SJC) [28 joints], patient's global assessment of disease activity [visual analog scale: 0=no disease activity to 100=maximum disease activity] and the erythrocyte sedimentation rate (ESR) for a total possible score of 2 to 10. DAS28 Remission is defined as a DAS28 score <2.6.
Time Frame: Week 24
Population: Participants from the Intent-to-treat population, all randomized participants who received study drug and had at least 1 post-baseline efficacy assessment, with data available at Baseline and Week 24. Last observation carried forward was used to impute missing tender and swollen joint counts. All other ACR components were used as observed.
Measure: Number; unit: Percentage of participants
Arm/Group | Adalimumab + Methotrexate | Tocilizumab + Methotrexate
Number analyzed (Participants) | 33 | 36
Percentage of participants | 30.3 | 36.1

2. Secondary Outcome: Percentage of Participants With American College of Rheumatology (ACR20) Response at Week 24
Description: ACR20 response is defined as a ≥ 20% improvement (reduction) compared with baseline for both total joint count-68 joints (TJC68) and swollen joint count-66 joints (SJC66), as well as for three of the additional five ACR core set variables: Patient's Assessment of Pain over the previous 24 hours: using a Visual Analog Scale (VAS) left end of the line 0=no pain to right end of the line 100=unbearable pain; Patient's Global Assessment of Disease Activity and Physician's Global Assessment of Disease Activity over the previous 24 hours using a VAS where left end of the line 0=no disease activity to right end of the line 100=maximum disease activity; Health Assessment Questionnaire: 20 questions, 8 components: dressing/grooming, arising, eating, walking, hygiene, reach, grip and activities, 0=without difficulty to 3=unable to do; and acute-phase reactant Erythrocyte Sedimentation Rate.
Time Frame: Baseline, Week 24
Population: Participants from the Intent-to-treat population, all randomized participants who received study drug and had at least 1 post-baseline efficacy assessment, with ACR score data available. Last observation carried forward was used to impute missing tender and swollen joint counts. All other ACR components were used as observed.
Measure: Number; unit: Percentage of participants
Arm/Group | Adalimumab + Methotrexate | Tocilizumab + Methotrexate
Number analyzed (Participants) | 33 | 35
Percentage of participants | 66.7 | 62.9

3. Secondary Outcome: Percentage of Participants With ACR50 Response at Week 24
Description: ACR50 response is defined as a ≥ 50% improvement (reduction) compared with baseline for both total joint count-68 joints (TJC68) and swollen joint count-66 joints (SJC66), as well as for three of the additional five ACR core set variables: Patient's Assessment of Pain over the previous 24 hours: using a Visual Analog Scale (VAS) left end of the line 0=no pain to right end of the line 100=unbearable pain; Patient's Global Assessment of Disease Activity and Physician's Global Assessment of Disease Activity over the previous 24 hours using a VAS where left end of the line 0=no disease activity to right end of the line 100=maximum disease activity; Health Assessment Questionnaire: 20 questions, 8 components: dressing/grooming, arising, eating, walking, hygiene, reach, grip and activities, 0=without difficulty to 3=unable to do; and acute-phase reactant Erythrocyte Sedimentation Rate.
Time Frame: Baseline, Week 24
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | Adalimumab + Methotrexate | Tocilizumab + Methotrexate
Number analyzed (Participants) | 33 | 35
Percentage of participants | 24.2 | 42.9

4. Secondary Outcome: Percentage of Participants With ACR70 Response at Week 24
Description: ACR70 response is defined as a ≥ 70% improvement (reduction) compared with baseline for both total joint count-68 joints (TJC68) and swollen joint count-66 joints (SJC66), as well as for three of the additional five ACR core set variables: Patient's Assessment of Pain over the previous 24 hours: using a Visual Analog Scale (VAS) left end of the line 0=no pain to right end of the line 100=unbearable pain; Patient's Global Assessment of Disease Activity and Physician's Global Assessment of Disease Activity over the previous 24 hours using a VAS where left end of the line 0=no disease activity to right end of the line 100=maximum disease activity; Health Assessment Questionnaire: 20 questions, 8 components: dressing/grooming, arising, eating, walking, hygiene, reach, grip and activities, 0=without difficulty to 3=unable to do; and acute-phase reactant Erythrocyte Sedimentation Rate.
Time Frame: Baseline, Week 24
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | Adalimumab + Methotrexate | Tocilizumab + Methotrexate
Number analyzed (Participants) | 33 | 35
Percentage of participants | 18.2 | 22.9

5. Secondary Outcome: Percentage of Participants With Good or Moderate European League Against Rheumatism (EULAR) DAS28 Responses at Week 24
Description: The DAS28 score is a measure of the subject's disease activity. It is based on the tender joint count (28 joints), swollen joint count (28 joints), patient's global assessment of disease activity (mm), and ESR. DAS28 total score ranges from 0 (best) to 10 (worst). A negative change from Baseline indicated improvement. European League Against Rheumatism (EULAR) Good response: DAS28 ≤ 3.2 or a change from Baseline < -1.2. EULAR Moderate response: DAS28 >3.2 to ≤ 5.1 or a change from Baseline < -0.6 to ≥ -1.2.
Time Frame: Baseline, Week 24
Population: Participants from the Intent-to-treat population, all randomized participants who received study drug and had at least 1 post-baseline efficacy assessment, with data available at Week 24. Last observation carried forward was used to impute missing tender and swollen joint counts. All other EULAR components were used as observed.
Measure: Number; unit: Percentage of participants
Arm/Group | Adalimumab + Methotrexate | Tocilizumab + Methotrexate
Number analyzed (Participants) | 33 | 36
Percentage of participants
  Moderate Response | 39.4 | 27.8
  Good Response | 30.3 | 58.3

6. Secondary Outcome: Percentage of Participants With DAS28 Low Disease Activity (LDAS) at Week 24
Description: The DAS28 score is a measure of the patient's disease activity calculated using the tender joint count (TJC) [28 joints], swollen joint count (SJC) [28 joints], patient's global assessment of disease activity [visual analog scale: 0=no disease activity to 100=maximum disease activity] and the erythrocyte sedimentation rate (ESR) for a total possible score of 2 to 10. LDAS is defined as DAS28 ≤3.2.
Time Frame: Week 24
Population: Participants from the Intent-to-treat population, all randomized participants who received study drug and had at least 1 post-baseline efficacy assessment, with data available at Baseline and Week 24. Last observation carried forward was used to impute missing tender and swollen joint counts. All other DAS28 components were used as observed.
Measure: Number; unit: Percentage of participants
Arm/Group | Adalimumab + Methotrexate | Tocilizumab + Methotrexate
Number analyzed (Participants) | 33 | 36
Percentage of participants | 30.3 | 58.3

7. Secondary Outcome: Change From Baseline in DAS28 Score at Week 24
Description: The DAS28 score is a measure of the patient's disease activity calculated using the tender joint count (TJC) [28 joints], swollen joint count (SJC) [28 joints], patient's global assessment of disease activity [visual analog scale: 0=no disease activity to 100=maximum disease activity] and the erythrocyte sedimentation rate (ESR) for a total possible score of 2 to 10. A higher value indicated higher disease activity. A negative change from Baseline indicated improvement.
Time Frame: Baseline, Week 24
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Adalimumab + Methotrexate | Tocilizumab + Methotrexate
Number analyzed (Participants) | 33 | 36
Score on a scale | -1.65 (1.541) | -2.80 (1.553)

8. Secondary Outcome: Change From Baseline in Swollen Joint Count (SJC) at Week 24
Description: 66 joints were assessed for swelling and joints are classified as swollen/not swollen giving a total possible swollen joint count score of 0 to 66. A negative change from Baseline indicated improvement.
Time Frame: Baseline, Week 24
Population: Intent-to-treat population included all randomized participants who received study drug and had at least 1 post-baseline efficacy assessment. Last observation was used to impute missing swollen joint counts.
Measure: Mean (Standard Deviation); unit: Joint count
Arm/Group | Adalimumab + Methotrexate | Tocilizumab + Methotrexate
Number analyzed (Participants) | 46 | 48
Joint count | -5.7 (7.56) | -11.3 (15.84)

9. Secondary Outcome: Change From Baseline in Tender Joint Count (TJC) at Week 24
Description: 68 joints are assessed for tenderness and joints are classified as tender/not tender giving a total possible tender joint count score of 0 to 68. A negative change from Baseline indicated improvement.
Time Frame: Baseline, Week 24
Population: Intent-to-treat population included all randomized participants who received study drug and had at least 1 post-baseline efficacy assessment. Last observation carried forward was used to impute missing tender joint counts.
Measure: Mean (Standard Deviation); unit: Joint count
Arm/Group | Adalimumab + Methotrexate | Tocilizumab + Methotrexate
Number analyzed (Participants) | 46 | 48
Joint count | -8.0 (14.62) | -13.9 (16.50)

10. Secondary Outcome: Change From Baseline in Patient Assessment of Pain Visual Analog Scale (VAS) at Week 24
Description: The patient assessed their pain using a 0 to 100 millimeter (mm) horizontal visual analogue scale (VAS). The left-hand extreme of the line equals 0 mm, and is described as "no pain" and the right-hand extreme equals 100 mm as "unbearable pain". A negative change from Baseline indicated improvement.
Time Frame: Baseline, Week 24
Population: Participants from the Intent-to-treat population, all randomized participants who received study drug and had at least 1 post-baseline efficacy assessment, with data available at Baseline and Week 24.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Adalimumab + Methotrexate | Tocilizumab + Methotrexate
Number analyzed (Participants) | 33 | 36
Score on a scale | -30.1 (20.57) | -23.8 (29.28)

11. Secondary Outcome: Change From Baseline in the Patient Global Assessment of Disease Activity VAS at Week 24
Description: The patient's global assessment of disease activity is assessed on a 0 to 100 millimeter (mm) horizontal visual analogue scale (VAS) by the patient. The left-hand extreme of the line equals 0 mm, and is described as "no disease activity" (symptom-free and no arthritis symptoms) and the right-hand extreme equals 100 mm, as "maximum disease activity" (maximum arthritis disease activity). A negative change from Baseline indicated improvement.
Time Frame: Baseline, Week 24
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Adalimumab + Methotrexate | Tocilizumab + Methotrexate
Number analyzed (Participants) | 33 | 36
Score on a scale | -30.2 (22.17) | -21.5 (28.89)

12. Secondary Outcome: Change From Baseline in the Physician Global Assessment of Disease Activity VAS at Week 24
Description: The physician global assessment of disease activity was assessed using a 0 to 100 mm horizontal visual analogue scale (VAS) by the physician. The left-hand extreme of the line equals 0 mm, and is described as "no disease activity" (symptom-free and no arthritis symptoms) and the right-hand extreme equals 100 mm, as "maximum disease activity" (maximum arthritis disease activity). A negative change from Baseline indicated improvement.
Time Frame: Baseline, Week 24
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Adalimumab + Methotrexate | Tocilizumab + Methotrexate
Number analyzed (Participants) | 33 | 36
Score on a scale | -37.0 (23.20) | -36.8 (32.34)

13. Secondary Outcome: Change From Baseline in High Sensitivity C-Reactive Protein (hsCRP) at Week 24
Description: Blood was collected for C-Reactive Protein (CRP) (a test for analysis of inflammatory and infectious disorders) and was analyzed at a central laboratory. The concentration of CRP was measured in milligram/liter (mg/L). A reduction in the level is considered an improvement
Time Frame: Baseline, Week 24
Population: Participants from the Intent-to-treat population, all randomized participants who received study drug and had at least 1 post-baseline efficacy assessment, with data available at Baseline and Week 24 for this outcome measure.
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Adalimumab + Methotrexate | Tocilizumab + Methotrexate
Number analyzed (Participants) | 33 | 35
mg/L | -1.127 (11.1261) | -7.474 (10.8446)

14. Secondary Outcome: Change From Baseline in Erythrocyte Sedimentation Rate (ESR) at Week 24
Description: Blood was collected for Erythrocyte Sedimentation Rate (ESR) (a test that assesses tissue inflammation) and was analyzed at a local laboratory. ESR was measured in millimeter/hour (mm/hr). A reduction in the level is considered an improvement.
Time Frame: Baseline, Week 24
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: mm/hr
Arm/Group | Adalimumab + Methotrexate | Tocilizumab + Methotrexate
Number analyzed (Participants) | 33 | 36
mm/hr | -1.2 (16.78) | -25.7 (25.52)

15. Secondary Outcome: Change From Baseline in Health Assessment Questionnaire-Disability Index (HAQ-DI) Score at Week 24
Description: The Stanford Health Assessment Questionnaire Disability Index (HAQ-DI) is a patient completed questionnaire specific for rheumatoid arthritis, consisting of 20 questions in 8 domains: dressing/grooming, arising, eating, walking, hygiene, reach, grip and common daily activities. There are 4 possible responses for each question: 0=without any difficulty, 1=with some difficulty, 2=with much difficulty and 3=unable to do. The score for each of the domains is the highest (worst) score in each domain. A patient must have a domain score for at least 6 of 8 domains to calculate a valid HAQ-DI score which is the sum of domain scores, divided by the number of domains that have a score for a total possible score minimum/maximum 0 (best) to 3 (worst). A negative change from Baseline indicated improvement.
Time Frame: Baseline, Week 24
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Adalimumab + Methotrexate | Tocilizumab + Methotrexate
Number analyzed (Participants) | 30 | 35
Score on a scale | -0.19 (0.437) | -0.36 (0.543)

16. Secondary Outcome: Change From Baseline in the Functional Assessment of Chronic Illness Therapy-Fatigue Scale (FACIT-Fatigue) Score at Week 24
Description: FACIT-F is a 13-item questionnaire. Patients scored each item on a 5-point scale: 0 (Not at all) to 4 (Very much). The larger the patient's response to the questions (with the exception of 2 negatively stated), the greater the patient's fatigue. For all questions, except for the 2 negatively stated ones, the code was reversed and a new score was calculated as (4 minus the patient's response). The sum of all responses resulted in the FACIT-Fatigue score for a total possible score of 0 (worse score) to 52 (better score). A higher score reflects an improvement in the patient's health status. A positive change from Baseline indicates improvement.
Time Frame: Baseline, Week 24
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Adalimumab + Methotrexate | Tocilizumab + Methotrexate
Number analyzed (Participants) | 32 | 34
Score on a scale | 5.6 (9.60) | 8.0 (9.33)

17. Secondary Outcome: Change From Baseline in Quality of Life Short Form (SF-36) Score at Week 24
Description: The SF-36 is a questionnaire used to assess physical functioning and is made up of eight domains: Physical Functioning, Role Physical, Bodily Pain, General Health, Vitality, Social Functioning, Role-Emotional and Mental Health. Transforming and standardizing these domains leads to the calculation of the Physical (PCS) and Mental (MCS) Component Summary measures. Scores ranging from 0 to 100, with 0=worst score (or quality of life) and 100=best score. A positive change from baseline indicates improvement.
Time Frame: Baseline, Week 24
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Adalimumab + Methotrexate | Tocilizumab + Methotrexate
Number analyzed (Participants) | 29 | 33
Score on a scale
  Physical Component Summary Score | 4.39 (6.110) | 5.84 (7.980)
  Mental Component Summary Score | 6.07 (12.171) | 6.84 (11.907)

18. Secondary Outcome: Change From Baseline in Routine Assessment of Patient Index Data 3 (RAPID3) Score at Week 24
Description: RAPID3 is a patient self reported assessment that combines the HAQ-DI [20 questions referring to 8 domains: dressing/grooming, arising, eating, walking, hygiene, reach, grip; common daily activities. Each domain has at least 2 component questions answered on a 4-point scale where 0=without any difficulty to 3=unable to do} converted to a score of 0-10, the Patients Assessment of Pain [Over the previous 24 hours: using a Visual Analog Scale (VAS) left end of the line 0=no pain to right end of the line 100=unbearable pain] converted to a score of 0-10 and the Patient's Global Assessment of Disease Activity [over the previous 24 hours using a VAS where left end of the line 0=no disease activity to right end of the line 100=maximum disease activity] converted to a score of 0-10. The 3 individual scales are summed for a raw score of 0-30 which is divided by 3 to achieve a total possible adjusted score of 0-10. A negative change from Baseline indicates improvement.
Time Frame: Baseline, Week 24
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Adalimumab + Methotrexate | Tocilizumab + Methotrexate
Number analyzed (Participants) | 30 | 35
Score on a scale | -2.17 (1.611) | -1.83 (2.257)

19. Secondary Outcome: Change From Baseline in Hemoglobin at Week 24
Description: Blood was collected at Baseline and Week 24. The samples were sent to a central laboratory for Hemoglobin analysis reported in gram/deciliter (g/dL). A positive number change from Baseline (a higher hemoglobin level compared to Baseline) indicated improvement
Time Frame: Baseline, Week 24
Population: Participants from the Intent-to-treat population, all randomized participants who received study drug and had at least 1 post-baseline efficacy assessment, with hemoglobin data available at Baseline and Week 24.
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Adalimumab + Methotrexate | Tocilizumab + Methotrexate
Number analyzed (Participants) | 32 | 35
g/dL | 1.2 (8.70) | 6.5 (12.01)

20. Secondary Outcome: Number of Participants With Serious Adverse Events (SAEs), Adverse Events (AEs), Discontinuation Due to AEs and Deaths
Description: An adverse event was considered any unfavorable and unintended sign, symptom, or disease associated with the use of the study drug, whether or not considered related to the study drug. Preexisting conditions that worsened during the study were reported as adverse events.
  A serious adverse event is any experience that suggests a significant hazard, contraindication, side effect or precaution that: results in death, is life-threatening, required in-patient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect or is medically significant.
Time Frame: 32 weeks
Population: Safety Population included all participants who received study drug and who had at least 1 post-dose safety assessment.
Measure: Number; unit: Participants
Arm/Group | Adalimumab + Methotrexate | Tocilizumab + Methotrexate
Number analyzed (Participants) | 48 | 48
Participants
  Any Adverse Event (AE) | 35 | 33
  Any Serious Adverse Event | 2 | 8
  AE leading to withdrawal | 3 | 5
  Death | 0 | 0

ADVERSE EVENTS:
Arm/Group | Adalimumab + Methotrexate | Tocilizumab + Methotrexate
Serious Adverse Events (participants affected / at risk) | 2/48 | 8/48
Other Adverse Events (participants affected / at risk) | 21/48 | 11/48
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Adalimumab + Methotrexate (N=48) | Tocilizumab + Methotrexate (N=48)
Pneumonia (Infections and infestations) | 1 | 1
Appendicitis (Infections and infestations) | 0 | 1
Bursitis infective (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 1
Hip fracture (Injury, poisoning and procedural complications) | 0 | 1
Tibia fracture (Injury, poisoning and procedural complications) | 0 | 1
Alanine aminotransferase increased (Investigations) | 1 | 0
Transaminases increased (Investigations) | 0 | 1
Ventricular tachycardia (Cardiac disorders) | 0 | 1
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Depression (Psychiatric disorders) | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Adalimumab + Methotrexate (N=48) | Tocilizumab + Methotrexate (N=48)
Upper respiratory tract infection (Infections and infestations) | 6 | 3
Nasopharyngitis (Infections and infestations) | 6 | 1
Bronchitis (Infections and infestations) | 3 | 2
Gastroenteritis (Infections and infestations) | 1 | 3
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 4 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 2 | 3
Headache (Nervous system disorders) | 1 | 3

LIMITATIONS AND CAVEATS:
Data interpretation was limited by the very small sample size (enrollment 1/7 of planned sample size; not powered for formal statistical analysis) and the open-label observation (study un-blinded following protocol amendment to terminate enrollment).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.